CLINICAL TRIAL: NCT01776970
Title: A Fase II, Randomized, Double-Blind, Placebo-Controlled, Multicentre Study for the Safety and Efficacy on Spasticity Symptoms of a Cannabis Sativa Extract in Motor Neuron Disease Patients
Brief Title: Safety and Efficacy on Spasticity Symptoms of a Cannabis Sativa Extract in Motor Neuron Disease
Acronym: CANALS
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ospedale San Raffaele (Other)
Collaborators: Fondazione Salvatore Maugeri (Other); Niguarda Hospital (Other); University of Padova (Other)
Responsible Party: Principal Investigator, Giancarlo Comi, Prof, Ospedale San Raffaele
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: CANALS
Record Dates: First submitted 2013-01-24; First posted 2013-01-28 (Estimated); Last update posted 2017-03-09 (Actual); Status verified 2017-03

CONDITIONS: Motor Neuron Disease; Amyotrophic Lateral Sclerosis (ALS)
Keywords: Motor Neuron Disease; Amyotrophic lateral sclerosis; Cannabinoids; Sativex; Spasticity
MeSH Terms: conditions — Motor Neuron Disease; Amyotrophic Lateral Sclerosis; Marijuana Abuse; Muscle Spasticity | interventions — nabiximols

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sativex (Experimental): Cannabis Sativa extract Oromucosal spray, containing THC (27 mg/ml):CBD (25 mg/ml)
  Interventions: Drug: Cannabis Sativa extract Oromucosal spray
- Placebo (Placebo Comparator): Placebo oromucosal spray
  Interventions: Drug: Cannabis Sativa extract Oromucosal spray

INTERVENTIONS:
Drug: Cannabis Sativa extract Oromucosal spray — Comparison between active drug (Cannabis Sativa extract Oromucosal spray, containing THC (27 mg/ml):CBD (25 mg/ml) vs placebo
  Other Names: Sativex

SUMMARY:
The clinical primary hypothesis is that there will be a difference between a Cannabis Sativa extract and placebo in their effect on spasticity in Motor Neuron Disease (MND) patients with signs of involvement of the upper motor neuron (UMN) resulting in disabling spasticity.

Secondary goals of the study are to evidence of improvement in other symptoms (in particular pain), and to show favourable trends on functionality measures. Finally, cannabis based drug safety and tolerability will be studied through vital parameters (including weight and pulmonary function) measurement, and analyzing ALS function rating scale progression slope hopefully, showing a slowing of the functional values decrease, owing to cannabis neuroprotective effects)

DETAILED DESCRIPTION:
CANALS project has as a main objective to analyse the safety profile, tolerability and efficacy of a Cannabis Sativa (Sativex) derivative on patients affected by spasticity due to motor neuron disease.

Muscular rigidity (or spasticity) is a symptom that affects many patients with motor neuron disease, concurring to reduce personal autonomy, patients' quality of life and can potentially cause secondary symptomatology (as pain or secondary muscular retractions). Currently available anti-spasticity drugs are often unsatisfactory and their pharmacological action can cause weakness as a secondary effect. There many arguments supporting the use of cannabinoid derivatives in motor neuron diseases. Cannabinoids receptor is expresses both in the brain and in the spinal cord. In animal models cannabinoids have an anti-spasticity effect. Moreover recent studies on ALS animal models demonstrated a neuroprotective effect of cannabinoids, including the preservation of the motor ability and a survival increase of the treated animals. Recently many clinical trials (some of them performed at the Neurological Division of San Raffaele Hospital) demonstrated cannabinoid efficacy on spasticity in Multiple Sclerosis patients. CAnnabinois would be able to reduce spasticity with no secondary weakness effect on treated patients. The results of these studies led to the drug approval in certain countries and by the European Community for the treatment of spasticity in Multiple Sclerosis.

The aim of this study is to analyze the safety, tolerability and efficacy profile of a Cannabis Sativa (Sativex) derivative on patients affected by spasticity due to motor neuron disease ( Amyotrophic Lateral Sclerosis and Primary Lateral Sclerosis). The study will be performed along 7 weeks. During the first week will be asked patients to note down in the clinical diary elements related to their symptomatology. Afterwards patients will be randomized in two groups: drug-treated and placebo treated. The study will be followed by a 6-weeks open-label phase during which all patients will receive the active drug (Phase B)

ELIGIBILITY:
Inclusion criteria:

Subjects must fulfil ALL of the following criteria:

* Written informed consent
* Subject able and willing to comply with all study requirements
* Affected by ALS, either of definite, probable or possible category according to the El Escorial revised criteria or by primary lateral sclerosis (Pringle's criteria)
* Affected of spasticity, equal or above 1 in the Ashworth Scale for spasticity in 2 or more muscle groups
* Who will judge spasticity a relevant cause of movements impairment
* Subject has spasticity due to MND of at least three months duration, which is not wholly relieved with current anti-spasticity therapy
* Subject fulfils at least one of the two criteria below. Subject must be either:

  1. Currently established on a regular dose of anti-spasticity therapy, or
  2. Previously tried and failed, or could not tolerate suitable anti-spasticity therapy
* Stabilization of factors affecting spasticity: any physiotherapy regimen or medication likely to affect spasticity will be optimised before the study and not altered in the 3 weeks before start of treatment
* Subject is willing for his or her name to be notified to the responsible authorities for participation in this study, as applicable.

Additional inclusion Criteria to be met at baseline

• Subjects have registered spasticity NRS scores via the personal clinical diary over the 6 days (day 2 to day 7) before randomization

Exclusion criteria:

* Any concomitant disease or disorder that has spasticity-like symptoms or that may influence the subject's level of spasticity
* Subjects receiving Botulinum Toxin during the preceding 6 months
* Bedridden and tracheotomised patients
* Fixed-tendon contractures
* Severe cognitive impairment
* Currently using or has used cannabis, cannabinoid-based medications or Acomplia (Rimonabant) within 30 days of study entry and unwilling to abstain for the duration of the study
* Any history or immediate family history of schizophrenia, other psychotic illness, severe personality disorder or other significant psychiatric disorder other than depression associated with their underlying condition
* Any known or suspected history of a diagnosed dependence disorder, current heavy alcohol consumption, current use of an illicit drug or current non-prescribed use of any prescription drug
* Subjects with poorly controlled epilepsy or recurrent seizures (Subjects who have had one or more fits in the year prior to Visit 1 will be excluded)
* Any known or suspected hypersensitivity to cannabinoids or any of the excipients
* Subject has experienced myocardial infarction or clinically relevant cardiac dysfunction within the last 12 months or has a cardiac disorder that, in the opinion of the investigator would put the subject at risk of a clinically relevant arrhythmia or myocardial infarction
* Subject has a diastolic blood pressure of <50 mmHg or >105 mmHg (when measured in a sitting position at rest for five minutes) or a postural drop in the systolic blood pressure of greater than 20 mmHg
* Personal history suggestive of relevant impaired renal or hepatic function
* Female subjects of child bearing potential, unless willing to ensure that they or their partner use effective contraception during the study and for three months thereafter
* Female subject who is pregnant, lactating or planning pregnancy during the course of the study and for three months thereafter
* Subjects who have received any IMP within the 8 weeks before Visit 1
* Any other significant disease or disorder which, in the opinion of the investigator, may either put the subject at risk because of participation in the study, or may influence the result of the study, or the subject's ability to participate in the study
* Unwilling to abstain from donation of blood during the study
* Patients will be asked not to drive while they will be receiving medication

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
modified 5 - points modified Ashworth scale (AS). | Week 7 (6 weeks after randomization)
  Improvement in the modified 5 - points modified Ashworth scale (AS). The variable for analysis will be the change in AS from the baseline (visit 2, Week 2) to the end of treatment (visit 4, Week 7).

SECONDARY OUTCOMES:
Mean weekly spasticity, spasm frequency and sleep disruption Numeric Rating Scale (NRS) score | Week 7 (6 weeks after randomizazion)
  Mean weekly spasticity, spasm frequency and sleep disruption NRS score at the end of treatment. The variable for analysis will be the change in mean NRS from the baseline (days 0-7) to the last week of treatment (usually days 42-49). Proportion of subjects completing the study and showing an improvement of 30% or more and 50% or more in NRS from Baseline (Week 1) and end of study (last seven days of treatment)

OTHER OUTCOMES:
Pain NRS score | Week 7 (6 weeks ater randomization)
  Pain will be measured with the mean of the last 3 days 0 - 10 daily pain intensity NRS.
Appetite increase | Week 7 (6 weeks after randomization)
  Weight difference before and at the end of the study.
Function (Ten meters walk test, ALS-FRS, Barthel ADL Index) | Week 7 (6 weeks aftar randomization)
  The time taken for the 10-metre walk, ALS-FRS and Barthel ADL Index will be analysed using the Visit 2 (week 1)result as baseline.
Global Impression of Change | Week 7 (6 weeks after randomization)
  Carer Global Impression of Change and ease of transfer Physician Global Impression of Change Subject Global Impression of Change
Safety | Week 4, week 7
  Adverse events, Vital Signs, Physical Examination , oral examination

CONTACTS AND LOCATIONS:
Overall Officials: Giancarlo Comi, MD, Principal Investigator — San Raffaele Scientific Institute
Locations (4):
- Italy (4):
  - San Raffaele Scientific Institute, Milan
  - Fondazione Salvatore Maugeri IRCCS, Istituto Scientifico, Milan
  - NEuroMuscular Omnicentre (NEMO), Fondazione Serena - H Cà granda, Milan
  - Universita' Degli Studi Di Padova, Azienda Ospedaliera Di Padova, Neurologic Department;, Padua

REFERENCES:
- [Derived] Riva N, Mora G, Soraru G, Lunetta C, Ferraro OE, Falzone Y, Leocani L, Fazio R, Comola M, Comi G; CANALS Study Group. Safety and efficacy of nabiximols on spasticity symptoms in patients with motor neuron disease (CANALS): a multicentre, double-blind, randomised, placebo-controlled, phase 2 trial. Lancet Neurol. 2019 Feb;18(2):155-164. doi: 10.1016/S1474-4422(18)30406-X. Epub 2018 Dec 13. PMID 30554828